CLINICAL TRIAL: NCT04008485
Title: Developing and Testing a Clinical Grade Magnetic Impedance Spectroscopy Device for Cervical Assessment to Predict Preterm Birth
Brief Title: Clinical Grade MIS Device for Cervical Assessment to Predict Preterm Birth
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sheffield Teaching Hospitals NHS Foundation Trust (Other)
Collaborators: University of Sheffield (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: STH19385
Record Dates: First submitted 2018-01-17; First posted 2019-07-05 (Actual); Last update posted 2023-11-18 (Actual); Status verified 2023-11

CONDITIONS: Preterm Birth
MeSH Terms: conditions — Premature Birth

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Asymptomatic high-risk women (Experimental): Women will be scheduled to attend for MIS measurement at 20-22 weeks, to be repeated at 26-28 weeks. This measurement will be taken at the same time as the routine examination which they receive when they attend the prematurity clinic. At each study visit the patient will undergo a vaginal examination. Triple high vaginal swabs will then be taken for bacteriology and fetal fibronectin. The sterile magnetic impedance probe will then be introduced, data being captured automatically by pressing the data capture button on the handle of the device. A transvaginal scan will also be performed to measure CL.
  Interventions: Device: Magnetic Electric Impedance Spectroscopy Device to predict PTB
- Symptomatic pregnant women (Experimental): These women (≥ 16 years of age) will be approached when they attend the labour delivery room or triage with symptoms of preterm labour as detailed above. As a matter of clinical routine these women receive a speculum examination, triple vaginal swabs taken, and fetal fibronectin and cervical length scans as indicated. The study will be explained to them and study materials provided. They will be asked to contact research staff by telephone or through their clinical midwife if they wish to participate. They will be given time to decide. If they agree to take part, written informed consent will then be obtained by research staff who will also conduct the MIS study. If clinical assessments have not already been performed by the time of obtaining consent they will be carried out at the same time
  Interventions: Device: Magnetic Electric Impedance Spectroscopy Device to predict PTB

INTERVENTIONS:
Device: Magnetic Electric Impedance Spectroscopy Device to predict PTB — During this phase, we will measure MIS in 100 women at high risk of PTB (Group 1) and 100 women with symptoms of PTB to confirm its predictive potential for PTB. To determine whether MIS assessment could prove a platform technique for other tests and treatments within existing antenatal care pathways for PTB, we will also assess vaginal swabs for fFN and measure cervical length (CL) by ultrasound.

SUMMARY:
Every year, globally, about 15 million babies are born preterm (before 37 weeks). This number is rising. Preterm birth (PTB) complications are the leading cause of death among children under 5 years of age, responsible for nearly 1 million deaths annually. PTB poses a strain on scarce health resources: each very premature baby costs tens of thousands of pounds in newborn care. One in 4 babies born before 28 weeks develop neurological impairment, a parent often having to give up work to care for an affected child. The prediction and prevention of PTB remain challenging because current methods, such as measuring the cervix by ultrasound, have limited accuracy. If a technique that reliably predicts PTB could be developed, there are care measures that can be employed to delay birth to reduce long-term disability/impairment. The Investigators have been studying whether they can detect the changes in cervical tissue structure and composition that precede PTB by using very low current Electrical Impedance Spectroscopy (EIS). Evidence recently showed that women at high risk of PTB (history of previous PTB), who deliver preterm, including delivery before 28 weeks gestation, have lower cervical "resistance" in mid-pregnancy than those who deliver at term. With NIHR funding, the investigators have developed a new device, based on a technique called magnetic impedance spectroscopy (MIS) that should address limitations of the EIS device for assessing PTB risk. The investigators now want to refine the new MIS device by minimising the signals it receives from other tissues around the cervix and making its measurements at internal body temperature more stable. The researchers also conduct clinical experiments to test whether it predicts PTB better than the previous EIS device, and check whether pregnant women find its use acceptable. This information will allow them to obtain UK regulatory approval to test the device in larger trials.

DETAILED DESCRIPTION:
The studies will be undertaken at the Jessop Wing (JW) Maternity Unit of the Royal Hallamshire Hospital, a tertiary referral unit with annual birth statistics of approximately 8000 births per annum. The JW receives in utero transfers from > 6 other hospitals in South Yorkshire and houses the regional neonatal intensive care unit with high dependency care facilities equipped to deal with extremely premature births, including those born at gestational ages borderline for viability (23-26weeks). The unit is therefore suited for the care of women at high risk of premature delivery and is well suited to house this study. The clinician on the core research team for this application also accepts referrals for high risk antenatal care and surveillance of women most at risk of premature delivery from colleagues in referring hospitals.

To reach this objective, the Investigators will package the project into three work packages (WP) with target milestones over 36 months. The time frames for the study phases are outlined below.

WP1. DURATION - 30 MONTHS, M1-30. LEAD J. HEALEY

Objectives:

* To recruit high-calibre research staff (Postdoctoral Research Associate Clinical Engineer and Clinical Research Fellow) at project initiation.
* To refine/optimise the hardware and software of the MIS device to enable a clinical grade version - the MIS Mark 2 device (in collaboration with Arrow Technical).
* To apply for MHRA regulatory approvals for a device that can be employed for follow-on multicentre studies, towards eventual CE Marking post-project.

Outline of work strands in WP1. Improvements on current MIS 1 device prototype that will be addressed during this work package (M1-M9) include the following:

1. Removal of measurement artefacts
2. Removal of probe handling sensitivity from perturbations of the electric field around the probe
3. Reduction in thermal drift by better choice of materials and coil assembly and the use of "mechanical chopping" of the magnetic field
4. Reduction of power dissipation in the probe in order to improve stability 5. Improving the ruggedness of the probe to cope consistently with clinical use 6. Fractionally reducing the probe diameter.

These will culminate in refinements to the device hardware and software (M8-9). The Investigators will also simultaneously consolidate the technical documentation, which have been systematically collected during the development of the MIS Mark 1 device (M1-M18), and submit an application to the MHRA for regulatory approvals by M19. Following iterations with the MHRA they anticipate obtaining final approvals by the MHRA by the end of this workpackage (M30).

PPI Input to WP1

* The Investigators will schedule their first PPI meeting in Month 3 - this meeting will include an induction programme for new PPI members, as well as a refresher session for current PPI members. The PPI group will deliberate on the research plan and the participant information leaflets and consent forms for the clinical studies that will be submitted for National Research Ethics Committee approvals.

  o This PPI meeting has successfully held on 27 April 2017
* A second PPI meeting in Month 11 will review project progress, consider the Mark 2 MIS device and advice on the planned submission to the MHRA.

WP1 Deliverables:

* Prompt initiation of project following successful pre-project employment of PDRA and Clinical Research Fellow.
* 1st PPI meeting Month 3.
* Manufacture of high-performance Mark 2 MIS cervical device by M10
* 2nd PPI meeting Month 11
* Submission of initial application for regulatory approvals by the MHRA by M19
* MHRA Regulatory approvals secured by M30 WP2. DURATION - 30 MONTHS, M 1- 30. LEAD PROF DILLY ANUMBA

Objectives:

During this phase, the Investigators will conduct clinical experimental studies to determine the predictive potential of the MIS Mark 2 device for preterm birth (PTB) in a cohort of asymptomatic women at risk of PTB (previous history of PTB, AHR) attending for pregnancy care (n=100), and another cohort of women (n=100) presenting to labour ward between 20-34 weeks with symptoms of preterm labour (regular uterine contractions - > 1 contraction every 10 minutes - but cervix less than 4 cm dilated, SYM). The rationale for sample size estimates is clarified later on this protocol.

Outline of work strands in WP2:

This WP will overlap with WP1 to ensure that technical project development occurs in tandem with the preparation for, and execution of, clinical experimental studies.

During this WP the Investigators will:

* Obtain research ethics and governance approvals (M1-M6).
* Generate preliminary data (M7-M18) that will be employed to: a) apply to the MHRA for regulatory approvals, and b) optimise the probe hardware and software further, and
* Conduct experimental studies on the cohorts detailed above (M8-M30) - recruit and study asymptomatic HR cohort (n=100) and symptomatic cohort (n=100) from M8 -M30 (22 months). In addition to standard care, the women will have an ultrasound scan to assess cervical length, vaginal swab specimen collection for fetal fibronectin determination and microbiological studies and MIS assessment at each of two study visits. Women with abnormal cervical cytology in the previous 3 years or with signs of ongoing cervical infection will be excluded from the studied.

Study conduct details:

• Target population and sample selection: Asymptomatic high-risk women. These participants (≥ 16 years of age) will have had no signs of cervical infection, no previous cervical surgery, and will have had a normal cervical smear within the previous 3 years. Prospective participants will be approached at their first hospital antenatal visit. The study will be explained and study materials provided. The participants will be asked to contact research staff by telephone or through their community midwife, or at the time of the participant's next attendance to the prematurity clinic or ultrasound scan appointment if the women wishes to participate. Written informed consent will then be obtained by research staff who will also conduct the two study visits. Women will be scheduled to attend for MIS measurement at 20-22 weeks, to be repeated at 26-28 weeks. This measurement will be taken at the same time as the routine examination which the participants receive when they attend the prematurity clinic. At each study visit the patient will undergo a vaginal examination. Triple high vaginal swabs will then be taken for bacteriology and fetal fibronectin. The sterile magnetic impedance probe will then be introduced, data being captured automatically by pressing the data capture button on the handle of the device. A transvaginal scan will also be performed to measure CL. The average duration of this assessment, from obtaining the swabs to completing the ultrasound scan, is about 7 minutes.

The above procedure will be carried out at each of the two study visits planned. Women attending the prematurity clinic are seen on average every two to three weeks. Consequently, cervical magnetic impedance spectroscopy measurements will not need to be measured at every hospital visit.

Symptomatic pregnant women. These women (≥ 16 years of age) will be approached when the participant attends the labour delivery room or triage with symptoms of preterm labour as detailed above. As a matter of clinical routine these women receive a speculum examination, triple vaginal swabs taken, and fetal fibronectin and cervical length scans as indicated. The study will be explained to them and study materials provided. The participants will be asked to contact research staff by telephone or through their clinical midwife if the participants wish to participate. The participant will be given time to decide. If the participant agrees to take part, written informed consent will then be obtained by research staff who will also conduct the MIS study. If clinical assessments have not already been performed by the time of obtaining consent the participant will be carried out at the same time

ELIGIBILITY:
Inclusion Criteria:

* ≥ 16 years of age
* no signs of cervical infection
* no previous cervical surgery
* had a normal cervical smear within the previous 3 years
* identified as asymptomatic high-risk antenatally (Asymptomatic high-risk women participants)
* Symptoms of preterm labour (Symptomatic Pregnant women participants)

Exclusion Criteria:

* < 16 years of age
* signs of cervical infection
* previous cervical surgery
* no cervical smear within previous 3 years
* not identified as symptomatic high-risk antenatally (Asymptomatic high-risk women participants)
* No symptoms of preterm labour (Symptomatic Pregnant women participants)

Min Age: 16 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 127 (Actual)
Dates: Start 2018-05-01 (Actual); Primary Completion 2021-06-29 (Actual); Study Completion 2021-10-31 (Actual)

PRIMARY OUTCOMES:
Cervical Resistivity | Week 20-22 of pregnancy
  Cervical resistivity measured by use of Magnetic Impedance Spectroscopy probe. Probe measurements will be compared against birth outcomes to determine predictive ability of probe for pre-term birth.
Cervical Resistivity | Week 26-28 of pregnancy
  Cervical resistivity measured by use of Magnetic Impedance Spectroscopy probe. Probe measurements will be compared against birth outcomes to determine predictive ability of probe for pre-term birth. Measuring changes from week 20-22 visit.

SECONDARY OUTCOMES:
Assess service-user acceptability of the MIS device | Within 1 month of week 26-28 visit
  Assess service-user acceptability of the MIS device for screening for preterm birth, previously confirmed to be good for EIS in qualitative studies using the Sheffield Mark V EIS device.
  Questionnaires administered to capture participant acceptability
Cost-effectiveness | At 24 months
  On the basis of our clinical observations update our previously-developed cost-effectiveness model of such a device for predicting PTB, and estimate the maximum price that allows the technology to be cost-effective using the "headroom" approach. All data to be captured and analysed by health economists at clinical trials unit.

CONTACTS AND LOCATIONS:
Overall Officials: Dilly OC Anumba, Prof, Principal Investigator — Honorary Consultant in Obstetrics and Gynaecology
Locations (1):
- Jessop Wing Hospital, Sheffield, South Yorkshire, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided